CLINICAL TRIAL: NCT04571879
Title: Nebulized Lidocaine and Intranasal Midazolam for Reducing Pain/Anxiety of Nasogastric Tube Insertion in Children: A Randomized Clinical Trial
Brief Title: Nebulized Lidocaine and Intranasal Midazolam for NGT Insertion in Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRC-01-19-442
Record Dates: First submitted 2020-09-10; First posted 2020-10-01 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2022-06

CONDITIONS: Procedural Anxiety; Procedural Pain
MeSH Terms: conditions — Pain, Procedural | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Nebulized 2% lidocaine hydrochloride 4 mg/kg to be delivered via nebulization (up to a maximum of 15 ml) and given over ½ hr.
  Intranasal midazolam 0.5 mg/kg delivered via intranasal atomization (up to a maximum of 10 mg).
  Interventions: Drug: Nebulized Lidocaine; Drug: Intranasal Midazolam
- Arm 2 (Experimental): Intranasal midazolam 0.5 mg/kg to be delivered via intranasal atomization (up to a maximum of 10 mg).
  Nebulized placebo (Normal saline) in a volume comparable to 2% lidocaine at 4 mg/kg (up to a maximum of 15 ml) and given over ½ hr.
  Interventions: Drug: Intranasal Midazolam
- Arm 3 (Placebo Comparator): Intranasal placebo (normal saline) in a volume comparable to midazolam 0.5 ml/kg to be delivered via intranasal atomization
  Nebulized placebo (Normal saline) in a volume comparable to 2% lidocaine at 4 mg/kg (up to a maximum of 15 ml) and given over ½ hr.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nebulized Lidocaine — Nebulized Lidocaine for Reducing Pain of Nasogastric Tube Insertion in Children
  Other Names: Nebulized Xylocaine
  Arms: Arm 1
Drug: Intranasal Midazolam — Intranasal Midazolam for reducing anxiety of Nasogastric Tube insertion
  Other Names: IN Midazolam
  Arms: Arm 1; Arm 2
Other: Placebo — Nebulized normal saline and intranasal normal sline
  Arms: Arm 3

SUMMARY:
Nasogastric tube (NGT) is a commonly performed procedure in the Emergency Department. Although it is not a major procedure, it is usually associated with a bad experience and cause discomfort and pain in kids. This randomized controlled double-blinded double-dummy trial aims to investigate the efficacy of local topical anesthetic and/or anxiolysis for pain/anxiety related to NGT insertion. Eligible patients are children with gastroenteritis aged 6 months to 5 years requiring NGT rehydration. The intervention are 3 arms of nebulized lidocaine with midazolam compared to nebulized midazolam alone or placebo. The primary outcome is procedure-related pain assessment using the Face, Legs, Activity, Cry, and Consolability (FLACC) scale during final NGT insertion attempt.

DETAILED DESCRIPTION:
Nasogastric tube (NGT) insertion is commonly performed in the emergency department (ED) which can cause some pain/anxiety [Shih S and Rosen P, 2018]. The pain/discomfort related to NGT insertion comes from anxiety, gagging and sensitivity of nasopharynx and oropharynx [Tapiawala SN et al, 2008]. Success rate depends on cooperation, which limits order for nasogastric tube insertion in most patients especially in non-pediatric hospitals.

The pain and anxiety associated with such procedures in kids is a source of noxious stimuli to the nervous system. Not only does pain have a negative impact on neurological development, but children whose pain has not been adequately treated in infancy or early childhood reported lower pain thresholds as adolescents and adults [Ruda M.A.et al, 2000]. If not addressed, this pain can lead to distress for children, their parents and those performing the procedures, preprocedural anxiety in the future and can result in negative long-term emotional outcomes [Blount R.L et al,2006; Brewer S.G. et al, 2006].

Nebulized 2% lidocaine at doses of 4 and 8 mg/kg has shown to be safe in infants and children, with all blood levels obtained were well below the toxic range [Gjonaj S et al, 1997]. Nebulized lidocaine in doses up to 8 mg/kg appears to be safe and gave statistically significant reduction in pain score when used before flexible bronchoscopy [Gjonaj S et al, 1997]. Nebulized/intranasal lidocaine did not seem to be of benefit when used alone in the two previous trials for NGT insertion in children [Babl FE et al,2009; Craig SS et al, 2019]. On the other hand it greatly reduced discomfort associated with NG tube in adult population [Cullen L et al, 2004]. This might be explained by the anxiety and lack of cooperation, especially in young kids, which might limit the validity of pain score during the whole procedure.

Midazolam has a controlled sedation with a quicker recovery time. The safety and tolerability profile of midazolam in pediatric patients is comparable/superior to that observed in adults [Pacifici GM, 2014]. Midazolam is a GABA receptor agonist providing anxiolysis for procedures in pediatric population. Midazolam has been shown to be safe and effective for use in children [Wilton NC et al,1988; Theroux MC et al, 1993]. Intranasal midazolam has shown improvements with anxiety and crying, as well as need for restraint [Theroux MC et al, 1993]. Midazolam anxiolysis has been tried in pediatrics and ordered as nebulization, found to have a plasma concentration bioavailability which is comparable to the intranasal midazolam by the ratio (nebulized:nasal) of 1:2.9. [McCormick AS et al, 2008]. Clinically effective serum concentrations of intranasal midazolam can be reached within less than 10 min after nasal application [Knoester PD et al, 2002].

Lidocaine / Midazolam has been commonly used in different procedures in pediatric emergency department; such as urethral catheterization, intravenous cannulation, lumbar puncture with a great safety margin.

ELIGIBILITY:
Inclusion Criteria:

1 Previously healthy children 6 months to 5 years old presenting with AGE and some dehydration who were planned to have a nasogastric tube inserted as part of their ED treatment.

Exclusion Criteria:

1. Indication for an urgent insertion of a nasogastric tube.
2. Congenital anomalies of nose, nasopharynx, oropharynx, or oral cavity.
3. .Patients allergic to midazolam or lidocaine.
4. .Congenital Heart disease or arrhythmia.
5. .Known hepatic or renal impairment
6. .Developmentally abnormal children
7. .Patients with seizure disorder
8. .Pre-existing abnormal neurological conditions
9. .Child is taking medications known to interact with lidocaine and/or midazolam (antiarrhythmic drugs, suxamethonium, phenytoin, antidepressants, propranolol, citicoline).
10. .Known case of severe gastroesophageal reflux disease or aspiration pneumonia.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Pain severity rating scale (FLACC) during insertion of NGT. | 1 year
  score from 0 to 10. Higher scores mean worse outcome

SECONDARY OUTCOMES:
Observer/caregiver pain severity rating: | 1 year
  Score from 1 to 100. Higher scores mean worse outcome
The ease of procedure: difficulty of insertion on an ordinal scale from 1 to 5, where 5 is the most difficult insertion. | 1 year
  Score from 1 to 5. Higher scores mean worse outcome
The number of attempts required to successfully insert the NGT | 1 year
  The number of attempts of successful NGT insertion
Procedural complications/adverse events. | 1 year
  Records complications and adverse effects
FLAC score at 30 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes and 180 minutes post insertion. | up to 180 minutes
  Scores from 0 to 10. Higher scores mean worse outcome
Length of stay in ED | up to 180 minutes
  Length of stay in minutes
Duration of NGT feed. | up to 180 minutes
  The observer records data on chart
Tolerated volume of NGT feed. | 1 year
  Amount of fluid (ml)

CONTACTS AND LOCATIONS:
Overall Officials: Fatihi Toaimah, MD, PhD, Principal Investigator — Hamad Medical Corporation
Locations (2):
- Qatar (2):
  - Pediatric Emergency Center, Hamad Medical Corporation, Doha
  - Sidra Medicine, Doha

REFERENCES:
- [Result] Shih S, Rosen P. Pain Management for Nasogastric Intubation in Pediatrics. Cureus. 2018 Oct 9;10(10):e3429. doi: 10.7759/cureus.3429. PMID 30555754
- [Result] Tapaiwala SN, Al Riyami D, Cole E. A painful and knotted nasogastric tube. CMAJ. 2008 Feb 26;178(5):568. doi: 10.1503/cmaj.070750. No abstract available. PMID 18299545
- [Result] Ruda MA, Ling QD, Hohmann AG, Peng YB, Tachibana T. Altered nociceptive neuronal circuits after neonatal peripheral inflammation. Science. 2000 Jul 28;289(5479):628-31. doi: 10.1126/science.289.5479.628. PMID 10915627
- [Result] Blount RL, Piira T, Cohen LL, Cheng PS. Pediatric procedural pain. Behav Modif. 2006 Jan;30(1):24-49. doi: 10.1177/0145445505282438. PMID 16330518
- [Result] Brewer S, Gleditsch SL, Syblik D, Tietjens ME, Vacik HW. Pediatric anxiety: child life intervention in day surgery. J Pediatr Nurs. 2006 Feb;21(1):13-22. doi: 10.1016/j.pedn.2005.06.004. PMID 16428010
- [Result] Gjonaj ST, Lowenthal DB, Dozor AJ. Nebulized lidocaine administered to infants and children undergoing flexible bronchoscopy. Chest. 1997 Dec;112(6):1665-9. doi: 10.1378/chest.112.6.1665. PMID 9404766
- [Result] Babl FE, Goldfinch C, Mandrawa C, Crellin D, O'Sullivan R, Donath S. Does nebulized lidocaine reduce the pain and distress of nasogastric tube insertion in young children? A randomized, double-blind, placebo-controlled trial. Pediatrics. 2009 Jun;123(6):1548-55. doi: 10.1542/peds.2008-1897. PMID 19482767
- [Result] Craig SS, Seith RW, Cheek JA, Wilson K, Egerton-Warburton D, Paul E, West A. Lidocaine and phenylephrine versus saline placebo nasal spray for the pain and distress of nasogastric tube insertion in young children and infants: a randomised, double-blind, controlled trial. Lancet Child Adolesc Health. 2019 Jun;3(6):391-397. doi: 10.1016/S2352-4642(19)30058-6. Epub 2019 Apr 15. PMID 31000379
- [Result] Cullen L, Taylor D, Taylor S, Chu K. Nebulized lidocaine decreases the discomfort of nasogastric tube insertion: a randomized, double-blind trial. Ann Emerg Med. 2004 Aug;44(2):131-7. doi: 10.1016/j.annemergmed.2004.03.033. PMID 15278085
- [Result] Pacifici GM. Clinical pharmacology of midazolam in neonates and children: effect of disease-a review. Int J Pediatr. 2014;2014:309342. doi: 10.1155/2014/309342. Epub 2014 Feb 18. PMID 24696691
- [Result] Wilton NC, Leigh J, Rosen DR, Pandit UA. Preanesthetic sedation of preschool children using intranasal midazolam. Anesthesiology. 1988 Dec;69(6):972-5. doi: 10.1097/00000542-198812000-00032. No abstract available. PMID 3195771
- [Result] Theroux MC, West DW, Corddry DH, Hyde PM, Bachrach SJ, Cronan KM, Kettrick RG. Efficacy of intranasal midazolam in facilitating suturing of lacerations in preschool children in the emergency department. Pediatrics. 1993 Mar;91(3):624-7. PMID 8441570
- [Result] McCormick AS, Thomas VL, Berry D, Thomas PW. Plasma concentrations and sedation scores after nebulized and intranasal midazolam in healthy volunteers. Br J Anaesth. 2008 May;100(5):631-6. doi: 10.1093/bja/aen072. Epub 2008 Apr 2. PMID 18385262
- [Result] Knoester PD, Jonker DM, Van Der Hoeven RT, Vermeij TA, Edelbroek PM, Brekelmans GJ, de Haan GJ. Pharmacokinetics and pharmacodynamics of midazolam administered as a concentrated intranasal spray. A study in healthy volunteers. Br J Clin Pharmacol. 2002 May;53(5):501-7. doi: 10.1046/j.1365-2125.2002.01588.x. PMID 11994056